CLINICAL TRIAL: NCT04311034
Title: A Phase Ib Study to Evaluate the Efficacy and Safety of RC48-ADC for Injection in Subjects With Advanced Non-small Cell Lung Cancer With HER2 Overexpression or HER2 Mutation
Brief Title: A Study of RC48-ADC in Subjects With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C004 NSCLC
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48 (Experimental)
  Interventions: Drug: RC48

INTERVENTIONS:
Drug: RC48 — Participants will be treated with RC48-ADC at a dose of 2.0 mg/kg, every 2 weeks. They will continue the medication until one of the following conditions occurred: disease progression, intolerance of toxicity, investigators believed that the subject could no longer benefit from treatment, or this study ended.

SUMMARY:
This study will evaluate the efficacy and safety of RC48-ADC for injection in subjects with advanced non-small cell lung cancer with HER2 overexpression or HER2 mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signed informed consent.
2. Male or female, Aged between 18 to 75 years.
3. Predicted survival ≥ 12 weeks.
4. According to UICC/AJCC 8th Edition, histologically and/or cytologically-confirmed, cannot be surgically removed, locally advanced or metastatic NSCLC.
5. Locally advanced or metastatic disease had failed at least one systemic treatment.
6. Based on imaging judgment (RECIST 1.1) or clinical status, tumor progression during or after the last treatment before enrollment.
7. HER2 protein overexpression (IHC 2+ or 3 +) or HER2 gene mutation (defined as exon 20 mutation), the previous test results confirmed by the researchers, both research centers and major research centers can be acceptable.
8. The researchers confirmed that the EGFR gene mutation status was negative or positive. For EGFR gene mutation-positive patients, one of the following is met: 1) T790M gene mutation negative, c-Met gene amplification negative and HER2 IHC 2+ or 3+ after first-generation EGFR-TKI drug resistance; 2) Third-generation EGFR-TKI treatment failed and HER2 IHC 2+ or 3+.
9. Measurable lesion according to the RECIST 1.1.
10. ECOG performance status score of 0 or 1.
11. Adequate organ function: LVEF ≥ 50 %. Hemoglobin ≥ 9g/dL; ANC ≥ 1.5×10^9 /L; Platelets ≥ 100×10^9 /L; Total bilirubin ≤ 1.5×ULN; ALT, AST and ALP ≤ 2.5×ULN and ≤ 5 x ULN with hepatic metastasis; Serum creatinine ≤1.5×ULN, or CrCl ≥ 60mL/min; INR≤ 1.5× ULN, APTT≤ 1.5× ULN.
12. For female subjects: should be surgically sterilized, postmenopausal, or agree to use a medically approved contraceptive (such as an intrauterine device, contraceptives, or condoms) during study treatment and within 6 months after the end of study, the blood pregnancy test within 7 days of study enrollment must be negative and must be non-lactating. Male subjects: Patients who should be surgically sterilized or agree to use a medically approved contraceptive during the study treatment period and within 6 months after the end of the study.
13. Willing and able to follow trial and follow-up procedures.

Exclusion Criteria:

1. Have used T-DM1 or participated in other HER2-ADC clinical studies.
2. Received anti-tumor treatment 4 weeks before study administration, including chemotherapy (late toxicity chemotherapy was 6 weeks before study administration), radiotherapy (palliative local radiotherapy for bone metastases was 2 weeks before the study administration), biological therapy (small molecule targeted drugs were 8 days before the study administration) or immunotherapy, etc.
3. Major surgery was performed within 4 weeks prior to study administration and did not fully recover.
4. Other clinical trial drugs have been used within 4 weeks before the start of study administration.
5. Live vaccine received within 4 weeks before the start of study administration.
6. Have received anti-tumor Chinese medicine treatment within 2 weeks before the start of study administration.
7. History of other malignant tumors within 5 years before signing the informed consent (except for non-melanoma skin cancer, cervical carcinoma in situ that has been effectively treated, or malignant tumors that have been resolved for more than 3 years after effective treatment and are considered to be cured) .
8. Toxicity of previous anti-tumor treatment has not recovered to CTCAE (version 4.03) 0-1, except for the following conditions: a. Hair loss; b. Pigmentation; c. Long-term toxicity caused by radiotherapy, which cannot be restored by the judgement of the investigator.
9. Active central nervous system (CNS) metastasis and/or cancerous meningitis (subjects who have received brain metastasis treatment can participate in this study, provided that the condition is stable (no evidence of progression confirmed by imaging studies at least 4 weeks before study dosing, and all neurological symptoms have returned to baseline levels), no evidence of new or enlarged brain metastases, and discontinuation of steroid treatment at least 7 days before the first dose of trial treatment. This exception does not include cancerous meningitis, which should be excluded whether clinical status was stable).
10. Diagnosed with HBsAg positive and HBV DNA positive, or HCV Ab positive, or HIV Ab positive.
11. Severe arterial/venous thrombosis or cardio-cerebral vascular accidents occurred within 1 year before the study, such as deep vein thrombosis, pulmonary embolism, cerebral infarction, cerebral hemorrhage, myocardial infarction, etc.
12. Active infections requiring systemic treatment.
13. Other lung diseases required systemic treatment such as active tuberculosis, interstitial lung disease, etc.
14. Uncontrolled systemic diseases such as diabetes, hypertension, cirrhosis, etc.
15. Heart failure graded 3 or above by the NYHA.
16. Pleural effusion, pericardial effusion, or peritoneal effusion with clinical symptoms that cannot be controlled by drainage or other methods.
17. Mental illness or substance abuse known to have an impact on compliance with study requirements.
18. Hypersensitivity or delayed allergic reaction to certain components of RC48-ADC or similar drugs.
19. Any other disease, metabolic abnormality, abnormal physical examination or abnormal laboratory test, etc., based on the judgment of the investigator, it is reasonable to suspect that the patient has a certain disease or condition unsuitable for the research drug, or will affect the interpretation of the research results, or putting patients at high risk.
20. Pregnant or lactating female or female / male who are planning to have children.
21. Insufficient adherence to participate in this clinical study.
22. Any other condition in which the investigator considers the patient unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate （ORR） | 15 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR).
Disease Control Rate (DCR) | 15 months
  Disease Control Rate (DCR) was defined as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents.
Progression Free Survival (PFS) | 15 months
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Duration of Response (DOR) | 15 months
  Duration of response is the length of time that a tumor continues to respond to treatment without the cancer growing or spreading.
Overall Survival (OS) | 24 months
  Overall survival, or OS, measures how long patients, who undergo a certain treatment regimen.

SECONDARY OUTCOMES:
Adverse events (AEs) | Up to 2 years
  The drug safety was assessed by investigator(s) according to NCI-CTCAE v4.03.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided